CLINICAL TRIAL: NCT05726435
Title: Effects of Soluble Dietary Fiber on Sport Efficiency and Fatigue Delay in Top Basketball Players
Acronym: FiberPlay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Antonio Starcevic, Associate professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IP-2016-06-3509
Record Dates: First submitted 2021-07-13; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Dietary Fiber; Sports; Sports Nutrition; Microbiota; Nutrition Surveys
Keywords: Fiber; Gastrointestinal Microbiota; Nutrition; 16S rRNA sequencing; Performance
MeSH Terms: interventions — NUTRIOSE; maltodextrin

STUDY DESIGN:
Intervention Model Description: Double-blind study of defined prebiotic supplementation for active basketball players investigating fiber effect on microbiota composition and delayed feeling of fatigue. There are two arms, active one receiving prebiotic fibre and control one receiving placebo. Each arm contains 7 randomly selected participants who signed informed consent and will receive supplementation during 4 weeks in total while being in the same training camp and under same training conditions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Program is used to make random selection and grouping of participants in two groups: experimental one receiving fiber and control one, receiving placebo. A research assistant who is not involved in study (neither design nor implementation) will pack prebiotic/placebo daily doses (20 grams/day) and provide nutritionist who is one of the investigators with doses for each participant. Only when the study is completed and all results processed will the information on who received fiber/placebo be released.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Seven randomly selected active basketball players will be supplemented with defined prebiotic fibre (20 grams per day divided in two 10 gram doses - 85% total fiber content) for the total duration of 4 weeks, while being stationed in the training camp under constant coach and nutrition expert surveillance.
  Interventions: Dietary Supplement: Soluble dietary fiber with prebiotic properties
- Control group (Placebo Comparator): Seven randomly selected active basketball players will be supplemented with placebo resembling prebiotic fibre in all visible and taste aspects (20 grams per day divided in two 10 gram doses) for the total duration of 4 weeks, while being stationed in the training camp under constant coach and nutrition expert surveillance.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soluble dietary fiber with prebiotic properties — 14 adult professional baskeyball players will be divided randomly in two groups, each containing 7 players. One group shall receive Nutriose fiber, two times per day 10 grams per dose in total duration of 4 weeks. Second group shall receive same amount of Placebo in form of Maltodextrin. Each group will undergo a series of sports performance tests and questionnaires and shall donate their feces several times during the study in order to monitor gut microbiota changes. The Nutriose group in this particular intervention contains 7 randomy selected players.
  Other Names: Nutriose
  Arms: Experimental group
Dietary Supplement: Placebo — 14 adult professional baskeyball players will be divided randomly in two groups, each containing 7 players. One group shall receive Nutriose fiber, two times per day 10 grams per dose in total duration of 4 weeks. Second group shall receive same amount of Placebo in form of Maltodextrin. Each group will undergo a series of sports performance tests and questionnaires and shall donate their feces several times during the study in order to monitor gut microbiota changes. This second (Placebo) group also consists of the 7 players and receives Maltodextrin supplementation. Since the study type is "double-blind", neither the participants (players) nor the person handing out the supplementation know the exact nature of fiber substance being handed during the entire duration of the trial. Independent statistician is handling the randomization of both interventions.
  Other Names: Maltodextrin
  Arms: Control group

SUMMARY:
Athlete nutrition is becoming an increasingly important factor on the path to achieving top results. Nutrients such as soluble fiber can alter the intestinal microbiota, resulting in metabolites with a positive effect on metabolism. Thus, the fibers become available, an additional source of energy to the host, have an anti-stress effect and delay the feeling of fatigue. The primary goal of the study is to determine the impact of soluble dietary fiber on increasing athletic efficiency, the secondary goal is to determine the impact of fiber on delaying fatigue. Subjects will be randomly divided into experimental and control group. The sample of variables will consist of genome microbiota genome sequencing data, measures to assess morphological characteristics, lower extremity explosive strength tests, and cardiovascular endurance. The statistical package SPSS will be used for data processing. The expected scientific contribution of this research is to expand the scientific knowledge about the importance of dietary fiber in the diet of athletes with the aim of improving sports performance.

DETAILED DESCRIPTION:
Material, participants, methodology and research plan The material will be soluble fiber NUTRIOSE and placebo. Nutriose, derived from corn, is generally well tolerated and no allergic reactions are known. Participants will be made aware of this in informed consent. If, however, there will be any adverse reactions in participant, participant will withdraw from the study immediately.

The participants will be 14 adult, professional basketball players. The sample of subjects was determined by the size of the group in the same training process in order to exclude the influence of different training processes on the research results. Participants who have used antibiotics in the last 3 months, participants with type 1 and 2 diabetes, and also who have used other ergogenic aids in the last 30 days and still using them are excluded.

Participants will be randomly divided into two groups: the experimental group that will consume the tested fibers and the control group that will consume placebo. Design is a double-blind study where an independent statistician will be entrusted with the randomization of subjects into the two groups.

Sample variables:

Methods: dietary methods, anthropometric methods, fatigue assessment questionnaire and fecal samples analysis.

The sample of variables consists of: fecal sample for intestinal microbiota sequencing, measures to assess morphological characteristics (body height, body weight, triceps skinfold, subscapular skinfold, chest skinfold, abdomen skinfold, suprailiocristal skinfold, thigh skinfold, axillary skinfold, fat percentage calculated by the seven skinfolds algorithm).

Dietary methods will be used to control eating habits and fiber intake prior to testing and to control diet during testing. The methods will be a food diary (three-day) and as an unannounced control of daily food intake once a week will be a 24-hour dietary recalls. The three-day food diary will show diet and average fiber intake just before the start of testing and unannounced control of daily food intake as evidence of unchanged eating habits during the study. All collected dietary data will be processed using Croatian food tables in addition to American tables for all foods whose chemical composition is not available in national tables.

In assessing the athletic performance of basketball players, emphasis will be placed on the explosive power of the lower extremities (concentric and eccentric contractions). Anthropometric methods will use tests to assess vertical explosive power (squat jump, countermovement jump, one legged countermovement jump, maximal countermovement jump, continuous jumps with straight egs, continuous jump with bent legs) with Optojump system and explosive power - sprint (5m, 10m and 20m sprint) with the Powertimer Newtest system. Aerobic endurance tests (BEEP test with sound signal) and anaerobic endurance test (300 m (15x20)) with Powertimer Newtest system will be used to assess cardiovascular endurance. Laboratory measurements will be performed within the Sports Diagnostic Center of the Faculty of Kinesiology, University of Zagreb.

Fecal samples will be collected at the Faculty of Food Technology and Biotechnology, University of Zagreb. Analysis of the composition of the intestinal microbiota by DNA sequencing from fecal samples will be performed using an Illumina NGS device.

Participants will complete a questionnaire on a daily basis in subjective feeling of fatigue on a scale of 1 to 10 (rate of perceived exertion).

Participants will have a daily short questionnaire on: bloating, change in stool consistency, nausea and weakness.

Research plan:

The research lasts a total of 8 weeks. Initial measurements before the start of supplementation include anthropometric testing and taking the first microbiota sample. This is followed by taking another microbiota sample 2 weeks after the start of supplementation. Final measurements follow at the end of 4 weeks of supplementation that include anthropometric testing and taking a third microbiota sample. Finally, the fourth microbiota sample will be 4 weeks after the final and 8 weeks after the initial measurements, respectively. After getting acquainted with the basics of testing, participants will sign a consent to participate.

Three days before the initial testing, participants will be explained how collect feces and the collection containers will be distributed. Each participant will be subjected to a dietary method of measuring food intake, a three-day diet diary and unannounced controls of daily food intake, once a week. Initial measurements will begin by collecting fecal-sampled containers. After measuring the morphological characteristics, tests to assess explosive power and aerobic and anaerobic capacities will be approached. After the initial testing, during the regular competition season, the participants of both groups will continue the training process without the possibility of additional training or changes in the training process. The experimental group (n = 7) will consume 2x8.5 g/day of soluble dietary fiber over four weeks, while the control group (n = 7) will consume the same amount of placebo carbohydrates. The dose was determined by previous studies with a proven effect on the morphological characteristics of participants and without side effects.

Participants will be taken by the respondents after the training in the presence of the research leader, and on the day off they will send a picture of an empty bag in mobile phone application. This will resolve "compliance." The training process will be the same for both groups, and participants will be advised not to change their diet pattern for two weeks prior to the test as well as for the duration of the experiment. After each training session and basketball game, respondents will complete a questionnaire in subjective feeling of fatigue on a scale of 1 to 10 (rate of perceived exertion). The final measurements are equal to the initial ones.

Data processing methods:

The sample size in the study was estimated through a test power of 70 % and a significance level of 5 %. The statistical program SPSS (Statistical Package for the Social Science), version 17.0., SPSS, Inc. will be used for data processing. Descriptive statistical parameters of the monitored variables will be calculated: arithmetic mean (AS), standard deviation (SD), minimum (MIN), maximum (MAX) and range result (RAS) and curvature (KURT) and distribution asymmetry (SKEW), and normality distribution by the Kolmogorov-Smirnov test. Multivariate and univariate analysis of variance (MANOVA and ANOVA) will be used to analyze the effects of training between initial and final measurements within groups, as well as to analyze differences in effects between groups. In case of statistically significant differences between groups, Tukey post hoc analysis will be used to determine the difference between specific groups. All conclusions will be drawn at the level of statistical error p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Professional basketball players from the same team participating in the same monitored training process

Exclusion Criteria:

* Diabetes or other chronic disease, taking sports performance enhancing drugs, taking antibiotics 3 months prior or during the course of the study

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Rapid microbiota change | 2 weeks
  The impact of fiber supplementation on gut microbiome shall assessed through monitoring of relative taxonomic abundance of bacteria that compose gut microbiota. DNA shall be extracted from collected faecal samples, stored at -80°C. DNA extraction shall be performed using the QIAamp® PowerFecal® DNA Kit. DNA concentration shall be quantified using Promega Quantus Flourometer before being sent to amplicon sequencing of variable regions 3 and 4 of the 16S rRNA gene with the primer set 341F (5'-CCTAYGGGRBGCASCAG -3') 806R (5'- GGACTACNNGGGTATCTAAT -3'). Obtained sequenceing raw data (reads) shall be analyzed using 'Quantitative Insights Into Microbial Ecology 2' (QIIME2) software in order to evaluate microbial composition of each sample. The comparison on intial sample (before intervention) and sample 1 (after 2 weeks) of supplementation shall provide a baseline insight into eventual rapid microbiota change as a response to supplementation/placebo.
Altered microbiota composition | 4 weeks
  Prolonged supplementation after initial 2 weeks will support the established altered gut microbiota in participants receiving fiber supplement. The impact of fiber supplementation on gut microbiome shall assessed through monitoring of relative taxonomic abundance of bacteria that compose gut microbiota. Gut microbiota DNA shall be extracted from collected faecal samples, stored at -80°C. DNA shall be processed in the same manner as previously described (Outcome 1). Obtained sequenceing raw data (reads) shall be analyzed using 'Quantitative Insights Into Microbial Ecology 2' (QIIME2) software in order to evaluate microbial composition of each sample. The comparison on intial sample (before intervention) and sample 2 (after 4 weeks) of supplementation shall provide an insight into eventual microbiota change as a response to prolonged supplementation/placebo.
Effect on the perception of fatigue | 4 weeks
  The major question is whether the moderately increasing fiber intake in athletes has the potential to support the intestinal microbiota and conversely positively impact training-induced perception of fatigue. In order to understand the impact of fiber consumption on the perception of fatigue, after each training session or match, the participants shall be asked to record and send a rating of perceived exertion through a mobile messaging application. The Borg's CR10 RPE scale shall be used for this purpose. This scale has a range from 0 to 10 (RPE - Rating of Perceived Exertion). The RPE scale is a tool used to monitor the perceptual response to training, as a method of determining physical exertion during exercise. The original RPE scale, developed more than 40 years ago, was primarily used to monitor aerobic load, but it still remains widely used in athlete tracking.

SECONDARY OUTCOMES:
Long-term microbiota impact | 8 weeks
  After total of 8 weeks fiber supplementation, one additional microbiota composition measurement (16S rRNA sequencing of donated fecal samples after 8 weeks of trial) will be taken after additional 4 weeks with no supplementation (intervention), in order to determine if the initial microbiota change caused by fiber supplementation can persist without additional fiber supplementation and to assess the potential for a long-term induced microbiota change. The comparison on intial sample (before intervention), sample 1 (after 2 weeks) of supplementation and sample 2 (after 4 weeks) with sample 3 (after 8 weeks) shall provide a baseline insight into microbiota change as a response to supplementation/placebo. DNA extraction and data processing shall be the same as in previous outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Starcevic, PhD, Principal Investigator — University of Zagreb, Faculty of Food Technology and Biotechnology
Locations (1):
- Faculty of Food Technology and Biotechnology, Zagreb, Croatia

REFERENCES:
- [Background] Wosinska L, Cotter PD, O'Sullivan O, Guinane C. The Potential Impact of Probiotics on the Gut Microbiome of Athletes. Nutrients. 2019 Sep 21;11(10):2270. doi: 10.3390/nu11102270. PMID 31546638
- [Background] Marttinen M, Ala-Jaakkola R, Laitila A, Lehtinen MJ. Gut Microbiota, Probiotics and Physical Performance in Athletes and Physically Active Individuals. Nutrients. 2020 Sep 25;12(10):2936. doi: 10.3390/nu12102936. PMID 32992765
- [Background] Clark A, Mach N. Exercise-induced stress behavior, gut-microbiota-brain axis and diet: a systematic review for athletes. J Int Soc Sports Nutr. 2016 Nov 24;13:43. doi: 10.1186/s12970-016-0155-6. eCollection 2016. PMID 27924137
- [Background] Mohr AE, Jager R, Carpenter KC, Kerksick CM, Purpura M, Townsend JR, West NP, Black K, Gleeson M, Pyne DB, Wells SD, Arent SM, Kreider RB, Campbell BI, Bannock L, Scheiman J, Wissent CJ, Pane M, Kalman DS, Pugh JN, Ortega-Santos CP, Ter Haar JA, Arciero PJ, Antonio J. The athletic gut microbiota. J Int Soc Sports Nutr. 2020 May 12;17(1):24. doi: 10.1186/s12970-020-00353-w. PMID 32398103
- [Background] Erdogan Z, Erdogan S, Aslantas O, Celik S. Effects of dietary supplementation of synbiotics and phytobiotics on performance, caecal coliform population and some oxidant/antioxidant parameters of broilers. J Anim Physiol Anim Nutr (Berl). 2010 Oct;94(5):e40-8. doi: 10.1111/j.1439-0396.2009.00973.x. PMID 20487099
- [Background] Lefranc-Millot C, Guerin-Deremaux L, Wils D, Neut C, Miller LE, Saniez-Degrave MH. Impact of a resistant dextrin on intestinal ecology: how altering the digestive ecosystem with NUTRIOSE(R), a soluble fibre with prebiotic properties, may be beneficial for health. J Int Med Res. 2012;40(1):211-24. doi: 10.1177/147323001204000122. PMID 22429361
- [Background] Farhangi MA, Javid AZ, Sarmadi B, Karimi P, Dehghan P. A randomized controlled trial on the efficacy of resistant dextrin, as functional food, in women with type 2 diabetes: Targeting the hypothalamic-pituitary-adrenal axis and immune system. Clin Nutr. 2018 Aug;37(4):1216-1223. doi: 10.1016/j.clnu.2017.06.005. Epub 2017 Jun 10. PMID 28669666
- [Background] Aliasgharzadeh A, Dehghan P, Gargari BP, Asghari-Jafarabadi M. Resistant dextrin, as a prebiotic, improves insulin resistance and inflammation in women with type 2 diabetes: a randomised controlled clinical trial. Br J Nutr. 2015 Jan 28;113(2):321-30. doi: 10.1017/S0007114514003675. PMID 27028002
- [Background] Li S, Guerin-Deremaux L, Pochat M, Wils D, Reifer C, Miller LE. NUTRIOSE dietary fiber supplementation improves insulin resistance and determinants of metabolic syndrome in overweight men: a double-blind, randomized, placebo-controlled study. Appl Physiol Nutr Metab. 2010 Dec;35(6):773-82. doi: 10.1139/H10-074. PMID 21164548
- [Background] Guerin-Deremaux L, Pochat M, Reifer C, Wils D, Cho S, Miller LE. The soluble fiber NUTRIOSE induces a dose-dependent beneficial impact on satiety over time in humans. Nutr Res. 2011 Sep;31(9):665-72. doi: 10.1016/j.nutres.2011.09.004. PMID 22024490
- [Background] Nazare JA, Sauvinet V, Normand S, Guerin-Deremaux L, Gabert L, Desage M, Wils D, Laville M. Impact of a resistant dextrin with a prolonged oxidation pattern on day-long ghrelin profile. J Am Coll Nutr. 2011 Feb;30(1):63-72. doi: 10.1080/07315724.2011.10719945. PMID 21697540